CLINICAL TRIAL: NCT00490867
Title: Effect of Long Term α-Lipoic Acid Treatment on Endothelial Function in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LipoicacidFBFV1.0
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2007-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alpha lipoic acid

SUMMARY:
In the present study, endothelium dependent vasodilation will be induced by administration of acetylcholine (ACh). To ascertain whether the vascular effects, if any, of α-lipoic acid are limited to the endothelium, endothelium independent vasodilation will also be assessed by administration of glyceroltrinitrate (GTN).

Study objectives To investigate the effect of α-lipoic acid therapy on endothelium dependent and independent vasodilation, assessed by forearm blood flow (FBF), in patients with type 2 diabetes mellitus

Study design

Randomized, double-blinded, parallel group study for 23 days:

Day 1: FBF responses to acetylcholine and glyceroltrinitrate Day 2-22: intravenous infusion of 600 mg α-lipoic acid or placebo Day 23: FBF responses to acetylcholine and glyceroltrinitrate

Study population 30 subjects with type 2 diabetes

Study medication Acetylcholine (ACh) - intraarterial infusion, 25, 50, 100 nmol/min, infusion period 3 minutes/dose level Glyceroltrinitrate (GTN) - intraarterial infusion, 4, 8, 16 nmol/min, infusion period 3 minutes/dose level α-lipoic acid - intravenous infusion of 600 mg in 250 ml saline solution over 30 minutes

Main outcome variables Forearm blood flow (Ratio between intervention and control arm) Additional outcome variables Arterial blood pressure, pulse rate, markers of inflammation and oxidative stress, Insulin plasma levels, Glucose plasma levels

Risk/benefit assessment The insertion of intravenous cannula may cause mild and transient pain. A minor hematoma may occur at the site of cannula insertion. The insertion of the intraarterial cannula is performed under local anaesthesia and causes mild pain. The meassurement of forearm bloodflow, espacialy the wrist cuff (>200 mmHG) may be uncomfortably. Local administration of drugs through a needle in the brachial artery allows the study of direct vascular effects of the drugs. Drug doses are 100 to 1000 times lower than a systemic effective dose, therefore no systemic adverse events are expected. There is experience in brachial artery infusions at our institution, and it is considered a safe technique. α-lipoic acid was well tolerated in healthy volunteers and subjects with diabetes at doses up to 600 mg intravenously and 1800 mg orally with side effects comparable with placebo. Altogether 50 ml blood will be collected throughout the study.

DETAILED DESCRIPTION:
Background

Type 2 (non-insulin-dependent) diabetes is associated with a marked increase in the risk of cardiovascular disease. Before overt cardiovascular disease occurs, impairment of vascular endothelial function is detectable. Endothelium-dependent vasodilation is impaired in patients with type 2 diabetes, indicating that diabetes is associated with endothelial dysfunction. Recently, formation of reactive oxygen species (ROS) has been linked to diabetes. These heterogeneous group of highly reactive compounds interact with NO and thereby inhibit vasodilation caused by NO. Formation of ROS is therefore thought to be an important mechanism by which type 2 diabetes induces endothelial dysfunction. α-Lipoic acid, which has been used for the treatment of diabetic neuropathy, was shown to have antioxidant capacities in vitro and animal experiments. Short term treatment with intraarterial α-lipoic acid was shown to improve endothelium dependent vasodilation in type 2 diabetics. However, to date, no data exists about the long term effcts of α-lipoic acid on vascular function in type 2 diabetics. In the present study, endothelium dependent vasodilation will be induced by administration of acetylcholine (ACh). To ascertain whether the vascular effects, if any, of α-lipoic acid are limited to the endothelium, endothelium independent vasodilation will also be assessed by administration of glyceroltrinitrate (GTN).

Study objectives To investigate the effect of α-lipoic acid therapy on endothelium dependent and independent vasodilation, assessed by forearm blood flow (FBF), in patients with type 2 diabetes mellitus

Study design

Randomized, double-blinded, parallel group study for 23 days:

Day 1: FBF responses to acetylcholine and glyceroltrinitrate Day 2-22: intravenous infusion of 600 mg α-lipoic acid or placebo Day 23: FBF responses to acetylcholine and glyceroltrinitrate

Study population 30 subjects with type 2 diabetes

Study medication Acetylcholine (ACh) - intraarterial infusion, 25, 50, 100 nmol/min, infusion period 3 minutes/dose level Glyceroltrinitrate (GTN) - intraarterial infusion, 4, 8, 16 nmol/min, infusion period 3 minutes/dose level α-lipoic acid - intravenous infusion of 600 mg in 250 ml saline solution over 30 minutes

Main outcome variables Forearm blood flow (Ratio between intervention and control arm) Additional outcome variables Arterial blood pressure, pulse rate, markers of inflammation and oxidative stress, Insulin plasma levels, Glucose plasma levels

Risk/benefit assessment The insertion of intravenous cannula may cause mild and transient pain. A minor hematoma may occur at the site of cannula insertion. The insertion of the intraarterial cannula is performed under local anaesthesia and causes mild pain. The meassurement of forearm bloodflow, espacialy the wrist cuff (>200 mmHG) may be uncomfortably. Local administration of drugs through a needle in the brachial artery allows the study of direct vascular effects of the drugs. Drug doses are 100 to 1000 times lower than a systemic effective dose, therefore no systemic adverse events are expected. There is experience in brachial artery infusions at our institution, and it is considered a safe technique. α-lipoic acid was well tolerated in healthy volunteers and subjects with diabetes at doses up to 600 mg intravenously and 1800 mg orally with side effects comparable with placebo. Altogether 50 ml blood will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetics; diagnosed on a clinical basis: positive family history; age of manifestation > 40 years; BMI >25; initial therapy without insulin
* Age: 40 - 65 years
* Body mass index between 26 and 35 [Wascher 1998]
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Treatment with concomitent therapy, including vasoactive drugs, is allowed during the study. Will not be changed during the study

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceeding the study
* History or signs of macrovascular disease
* History of hypertensitivity to the trial drug or to drugs with a similar chemical structure
* Changes in concomitant therapy during the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Clinical Pharmacology - Medical University Vienna